CLINICAL TRIAL: NCT05947370
Title: The Effect of Berberine on the Secretion of Incretin in Normal Man
Brief Title: Berberine on the Secretion of Incretin
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Jin-Kui Yang, professor, Beijing Tongren Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BBR incretin
Record Dates: First submitted 2023-06-04; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Berberine Chloride (Experimental): This study employed a randomized, double-blind, placebo-controlled, two-period crossover design: subjects were randomized into two groups of equal size. The random allocation was conducted by asking volunteers to select the randomized number generated by computer. Each number represented placebo or BBR, and each group has the same number of numbers. The dosing sequence in the first group was oral BBR in the first cycle and oral placebo in the second cycle. The second group was administered placebo in the first cycle and BBR in the second cycle. Take the second dose 14 days after the first dose. After the last dose, continue to observe for 14 days to watch for side effects. On each experimental day, after an overnight fast, the subjects received a single oral dose of 1 g of BBR or a corresponding dose of the placebo.
  Interventions: Drug: Berberine Chloride; Drug: Placebo
- Placebo control (Placebo Comparator): This study employed a randomized, double-blind, placebo-controlled, two-period crossover design: subjects were randomized into two groups of equal size. The random allocation was conducted by asking volunteers to select the randomized number generated by computer. Each number represented placebo or BBR, and each group has the same number of numbers. The dosing sequence in the first group was oral BBR in the first cycle and oral placebo in the second cycle. The second group was administered placebo in the first cycle and BBR in the second cycle. Take the second dose 14 days after the first dose. After the last dose, continue to observe for 14 days to watch for side effects. On each experimental day, after an overnight fast, the subjects received a single oral dose of 1 g of BBR or a corresponding dose of the placebo.
  Interventions: Drug: Berberine Chloride; Drug: Placebo

INTERVENTIONS:
Drug: Berberine Chloride — Traditional Chinese medicine
Drug: Placebo — Placebo control

SUMMARY:
Berberine (BBR) is the main active ingredient of the ancient Chinese herb medicine Coptis. The hypoglycemic effect of BBR has been demonstrated in numerous studies. Although BBR is safe and effective in the treatment of diabetes, its exact hypoglycemic mechanism is still unclear. Jin-Kui Yang found that BBR can promote GLP-1 secretion from intestinal L cells in mice in vitro and in vivo, thereby achieving the effect of lowering blood glucose, but it is still unknown whether BBR can promote incretin secretion in humans. In this study, investigators plan to examine the effect of BBR on secretion of incretin in human.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in the trial and signed informed consent form.
2. Healthy male subjects aged 18-45 years (including 18 and 45 years).
3. No history of current or former diseases such as heart, liver, kidney, gastrointestinal tract, nervous system, respiratory system, mental disorders and metabolic abnormalities that the investigator considers meaningful; no physical examination, electrocardiogram, and laboratory examination results abnormality or abnormality has no clinical significance (subject to the judgment of the physician).
4. Body mass index of 18.0-25.0 kg/cm2 (including 18.0 and 25.0 kg/cm2) and no centripetal obesity (waist-to-hip ratio less than 0.9).
5. No family history of diabetes mellitus and obesity.
6. Normal glucose tolerance (fasting blood glucose <6.1 mmol/L and 2h blood glucose <7.8mmol/L after oral administration of 75g glucose) and normal insulin secretion function (as judged by the investigator through the results of insulin release experiment).
7. Able to communicate well with the investigator and complete the study in accordance with the study regulations.

Exclusion Criteria:

1. Infection with hepatitis (A, B, or C), HIV and syphilis.
2. Those with clear allergy to berberine hydrochloride or its preparation components; those with drug (including salicylic acid) allergy, history of allergic diseases or allergic constitution.
3. Patients with hemolytic anemia and glucose-6-phosphate dehydrogenase deficiency.
4. Those who have used any prescription medication, herbal medicine within 4 weeks prior to dosing and/or taken over-the-counter medication (except for subjects with occasional or restricted use of paracetamol), supplements (except for routine vitamin supplementation) within 2 weeks prior to dosing.
5. Cumulative amount of blood loss (eg. blood donation) over 400mL within 3 months prior to baseline visit and during the study.
6. Heavy smokers (25 or more cigarettes per day) and heavy drinkers (14 units of alcohol per week, 1 unit = 285ml of beer, or 25ml of spirits, or 100ml of wine).
7. Those with a history of substance abuse or positive urine test for prohibited drugs.
8. Those who participated in any clinical trial within 1 month prior to the trial, or those who plan to participate in other clinical trials during or within 1 month after the end of the trial.
9. Other circumstances that the investigator considers unsuitable for participation in this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Differences of serum GLP-1 levels between BBR and placebo treatment groups during the glucose tolerance test. | 4 hours
  To compare the mean serum GLP-1 in the two groups during glucose tolerance test.
Differences of serum GIP levels between BBR and placebo treatment groups during the glucose tolerance test. | 4 hours
  To compare the mean serum GIP levels in the two groups during glucose tolerance test.
Differences of blood glucose levels between BBR and placebo treatment groups during the glucose tolerance test. | 4 hours
  To compare the mean blood glucose levels in the two groups during glucose tolerance test.

SECONDARY OUTCOMES:
Differences of serum insulin levels between BBR and placebo treatment groups during the glucose tolerance test. | The time frame is the same as Primary Outcome Measure 1
  To compare the mean insulin levels in the two groups during glucose tolerance test.
Differences of serum C-peptide levels between BBR and placebo treatment groups during the glucose tolerance test. | 4 hours
  To compare the mean serum C-peptide levels in the two groups during glucose tolerance test.
Differences of serum potassium levels between BBR and placebo treatment groups during the glucose tolerance test. | 4 hours
  To compare the mean serum potassium levels in the two groups during glucose tolerance test.
Differences of serum sodium levels between BBR and placebo treatment groups during the glucose tolerance test. | 4 hours
  To compare the mean serum sodium levels in the two groups during glucose tolerance test.
Differences of serum chloride levels between BBR and placebo treatment groups during the glucose tolerance test. | 4 hours
  To compare the mean serum chloride levels in the two groups during glucose tolerance test.
Differences of serum calcium levels between BBR and placebo treatment groups during the glucose tolerance test. | 4 hours
  To compare the mean serum calcium levels in the two groups during glucose tolerance test.

OTHER OUTCOMES:
Differences of heart rate between BBR and placebo treatment groups during the glucose tolerance test. | 4 hours
  To compare the mean heart rate in the two groups during glucose tolerance test.
Differences of QT-interval duration between BBR and placebo treatment groups during the glucose tolerance test. | 4 hours
  To compare the mean QT-interval duration in the two groups during glucose tolerance test.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Hao Wang, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lan J, Zhao Y, Dong F, Yan Z, Zheng W, Fan J, Sun G. Meta-analysis of the effect and safety of berberine in the treatment of type 2 diabetes mellitus, hyperlipemia and hypertension. J Ethnopharmacol. 2015 Feb 23;161:69-81. doi: 10.1016/j.jep.2014.09.049. Epub 2014 Dec 10. PMID 25498346
- [Background] Luthra A, Misra A. The marketing of unproven drugs for diabetes and dyslipidaemia in India. Lancet Diabetes Endocrinol. 2015 Oct;3(10):758-60. doi: 10.1016/S2213-8587(15)00328-9. No abstract available. PMID 26386988